CLINICAL TRIAL: NCT01671748
Title: Pragmatic Randomised Controlled Trial of MIST Ultrasound Therapy Compared to UK Standard Care for the Treatment of Non-healing Venous Leg Ulcers.
Brief Title: MIST Ultrasound Therapy Compared to United Kingdom Standard Care for the Treatment of Non-healing Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Celleration, Inc. (Industry)
Responsible Party: Principal Investigator, Professor Keith G Harding, Director - Institute for Translation, Innovation, Methodology and Engagement (TIME), Cardiff University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-SUR-5323
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-07

CONDITIONS: Varicose Ulcer
Keywords: Venous Leg Ulcer; Varicose Ulcer; Chronic ulcer; Chronic wound; Ultrasound therapy; MIST device; Wound healing; Low frequency non contact ultrasound
MeSH Terms: conditions — Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Active Comparator): Standard treatment for VLUs is administered once a week, i.e. compression bandaging and non-adherent dressing, with debridement if required.
  Interventions: Other: Standard Care
- MIST and Standard Care (Experimental): MIST ultrasound therapy is applied for between 3 and 12 minutes (depending on wound size) 3 times a week in combination with standard treatment for VLUs of compression bandaging and non-adherent dressing change 3 times a week, with debridement as required.
  Interventions: Device: MIST ultrasound therapy; Other: Standard Care

INTERVENTIONS:
Device: MIST ultrasound therapy — Low frequency, non-contact ultrasound system delivering therapeutic ultrasound via a fine saline mist to the wound bed.
  Other Names: MIST non-contact low-frequecy ultrasound device; MIST
  Arms: MIST and Standard Care
Other: Standard Care — Compression bandaging, non-adherent dressing, and debridement if required.

SUMMARY:
Chronic venous leg ulcers (VLUs) impact negatively on patients' quality of life. Standard treatment in the UK for patients with VLUs is compression bandaging or stockings. The MIST ultrasound system is a noncontact device which delivers low frequency ultrasound through a gentle saline mist directed at a patient's wound. This study aims to determine whether the use of the MIST device used in combination with standard treatments can improve healing of VLUs compared to UK standard practice. This will be assessed by measuring any reduction in wound size in the two groups after receiving 8 weeks of either Standard Care once a week or MIST combined with Standard Care three times a week.

DETAILED DESCRIPTION:
Venous leg ulcers (VLUs) are wounds which are often chronic and difficult to heal. VLUs affect between 1 and 3.2 people per 1000; they cause pain, reduced mobility and impact negatively on patients' quality of life (QoL). Standard treatment for patients with VLUs is the application of strong, sustained compression with bandages or stockings. This pragmatically-designed study aims to determine whether the use of a device called MIST used in combination with standard treatments can improve healing of VLUs compared to UK standard practice. It will also show whether the MIST regimen improves participants' QoL and reduces the incidence of infection.

The MIST ultrasound system is a non-contact device which delivers low-frequency ultrasound through a gentle saline mist directed at a patient's wound. Patients (over 18 years old) will be invited to take part in this study if they have had a VLU for 6 weeks or more, which measures between 5 and 100 cm^2, and is not infected. Participants with diabetes must show good blood glucose control, and those with underlying chronic disorders which may affect wound healing will be excluded.

All study participants will receive four weeks of standard treatment once a week at a single clinic at the Wound Healing Research Unit (WHRU), University Hospital of Wales. Patients whose wounds reduce by more than 40% during this time will be withdrawn from the study. Remaining patients will be randomly allocated to either the active group or the control group to receive a further eight weeks of treatment. Participants in the active group will receive treatment with the MIST device three times a week, as well as standard care (change of compression bandage and dressings) three times a week. The control group will receive UK standard care (which is dressing and compression bandage change at least once a week). The participants' ulcers will be measured and photographed once a week, and the wound characteristics will be assessed. Changes in participants' health related QoL will be assessed using a questionnaire at the beginning and end of the trial. Wound recurrence rates 90 days after the end of the treatment will be assessed by telephoning patients.

ELIGIBILITY:
Inclusion Criteria:

* Venous leg ulcers (as diagnosed by the clinician)
* Ankle Brachial Pressure Index (ABPI) >0.8
* If multiple ulcers are present treat largest ulcer only (index ulcer) with minimum distance of 1 cm between index ulcer and any other ulcer
* 18 years or older
* Ulcer size of 5 cm^2 - 100 cm^2 (with no longest length being greater than 10 cm) at randomisation point (week 5)
* Mobile enough to attend clinic
* Index ulcer between 6 weeks and 5 years duration prior to screening date

Exclusion Criteria:

* Uncontrolled diabetes (Hba1c ≥12%) as tested within the past 3 months
* Index ulcer has active infection on day of inclusion requiring use or oral or IV antibiotics
* Renal failure
* Index ulcer has exposed tendons, ligaments, muscle, or bone
* Osteomyelitis or cellulitis or gangrene in study limb
* Subjects with amputation above a trans metatarsal amputation (TMA) in the study limb
* Subjects with active malignancy on the study limb
* Index ulcer that is of arterial disease aetiology
* Females of child bearing potential who are not willing to use a method of highly effective contraception during the entire study
* Planned vascular surgery, angioplasty, or thrombolysis procedures within the study period, or 6 weeks post-operatively
* Planned surgical procedure during the study period for the index wound
* Prior skin replacement, negative pressure therapy, ultrasound therapy applied to the index wound 2 weeks before screening
* Oral or IV antibiotics within 48 hours of baseline measurements
* Growth factor therapy within previous 14 days of screening date
* Currently receiving or has received radiation or chemotherapy within 3 months of randomisation
* Pregnant or breast feeding women
* Subject is currently enrolled or has been enrolled in the last 30 days in another investigational device or drug trial
* Subject's wound would require ultrasound near an electronic implant or prosthesis
* Subjects lacking capacity to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith G Harding, Professor, Principal Investigator — Wound Healing Research Unit, Cardiff University
Locations (1):
- Wound Healing Research Unit, Cardiff University, Cardiff, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study procedures took place in a single dedicated unit specialising in wound healing research, between August 2012 and November 2013.
Pre-assignment Details: All enrolled patients received 4 weeks of SOC prior to random allocation (run-in phase). Patients whose wounds reduced by >40% in the first 4 weeks were withdrawn and did not progress to random allocation.
Groups:
- Standard of Care: Standard of Care (SOC) was compression bandaging and non-adherent dressing at least once a week (more frequent visits if clinically necessary). Debridement was performed as required.
- NLFU and Standard of Care: Non-contact low frequency ultrasound (NLFU) using MIST ultrasound therapy is applied for between 3 and 12 minutes (depending on wound size) 3 times a week in combination with standard treatment for VLUs of compression bandaging and non-adherent dressing change 3 times a week, with debridement as required.
Period: 4 Week run-in Phase
Arm/Group | Standard of Care | NLFU and Standard of Care
Started | 47 | 0
Completed | 36 | 0
Not Completed | 11 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Not eligible | 9 | 0
Period: 12 Week Treatment Phase
Arm/Group | Standard of Care | NLFU and Standard of Care
Started | 19 | 17
Completed | 19 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | NLFU and Standard of Care | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (12.2) | 70.5 (12.7) | 69 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19 | 17 | 36
History of leg ulceration (months) [Mean (Standard Deviation); unit: months] | 94.7 (83.2) | 109.7 (112.2) | 101.8 (96.8)
Index ulcer duration (months) [Mean (Standard Deviation); unit: months] | 22.3 (18.5) | 15.7 (12.0) | 19 (16)
Wound size at enrolment (cm^2) [Mean (Standard Deviation); unit: cm^2] | 19.4 (14.9) | 15.9 (9.9) | 17.8 (12.7)
Change in wound size during run-in phase (%) [Mean (Standard Deviation); unit: percentage change in wound area] | -13.0 (25.2) | -10.9 (23.9) | -12.0 (24.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Wound Area
Description: Wound area is measured weekly using a digital wound imaging device. The wound boundary is digitally traced by a blinded assessor. Percentage and actual change in wound area between start of treatment (week 5) and end of treatment (week 13) is evaluated.
Time Frame: Week 5 to 13
Population: All patients included in the analysis; Intention to treat (ITT); Values have been adjusted for the influence of the covariate (wound area at the start of treatment)
Measure: Mean (Standard Deviation); unit: percentage change in wound area
Arm/Group | Standard of Care | NLFU and Standard of Care
Number analyzed (Participants) | 19 | 17
percentage change in wound area | -39.2 (38.0) | -46.6 (38.1)
Statistical Analysis 1: Comparison: Standard of Care vs NLFU and Standard of Care; The study was powered to detect a difference in the change in wound area of 20% between the two arms with a two sided significance level and power of 90%. A standard deviation of 17.5% came from published literature. A minimum of 17 patients in each arm was required; Test type: Superiority or Other; p = 0.565, ANCOVA — ANCOVA was used to analyse differences between the NLFU+SOC and SOC arms of the primary endpoint, percentage change in wound area from baseline (week 5) to final visit (week 13). Patients' baseline (week 5) wound area was used as the covariate; Mean Difference (Final Values) = -7.4, 95% CI 2-sided [-33.4 to 18.6]

2. Secondary Outcome: Change in Overall Health Related Quality of Life (HRQoL) From Week 1 (Start) and Week 13 (Exit)
Description: On the first and final visit participants were invited to complete a Cardiff Wound Impact Schedule (CWIS) a validated questionnaire designed to measure the impact of chronic wounds on patient health-related quality of life (HRQoL). The overall HRQoL question asks patients to rate their overall quality of life over the past week by circling a number between 0 and 10. Low scores indicate poor quality of life, and high score indicate good quality of life. Change in HRQoL was calculated by subtracting week 1 values from week 13 values.
  CWIS has been validated in the following paper: Price and Harding (2004) The Cardiff Wound Impact Schedule: the development of a condition specific questionnaire to assess health-related quality of life in patients with chronic wounds. International Wound Journal 1(1):10-17
Time Frame: Week 1 (start) and week 13 (exit)
Population: All patients were analysed by ITT
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | NLFU and Standard of Care
Number analyzed (Participants) | 19 | 17
units on a scale | 0 [-1 to 1] | -1 [-2 to 2]
Statistical Analysis 1: Comparison: Standard of Care vs NLFU and Standard of Care; ANCOVA was used for change in HRQoL from week 1 to week 13 (with week 1 HRQoL score as the covariate); Test type: Superiority or Other; p = 0.490, ANCOVA

3. Secondary Outcome: Change in Ulcer Pain Between Week 5 (Randomisation) and Week 13 (Exit)
Description: Pain was scored by each patient on a visual analogue score (VAS) from 0 to 100. A VAS score of 0 indicated no pain whilst a VAS score of 100 indicated worst possible pain. Change in pain scores were calculated by subtracting week 5 values from week 13 values.
Time Frame: Weeks 5 to 13
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Standard of Care | NLFU and Standard of Care
Number analyzed (Participants) | 19 | 17
scores on a scale | -5.27 (14.84) | -14.35 (14.85)
Statistical Analysis 1: Comparison: Standard of Care vs NLFU and Standard of Care; ANCOVA was used for change in pain score (VAS) from week 5 to week 13 (covariate was baseline pain score); Test type: Superiority or Other; p = 0.078, ANCOVA; Mean Difference (Net) = -9.08, 95% CI 2-sided [-19.23 to 1.06]

4. Secondary Outcome: Incidence of Wound Infection
Description: Median number of wound infections per patient (as demonstrated by clinical symptoms) from beginning of treatment (week 5) and end of treatment (week 13).
Time Frame: Weeks 5 to 13
Population: All patients included; ITT.
Measure: Median (Inter-Quartile Range); unit: Number of infections per patient
Arm/Group | Standard of Care | NLFU and Standard of Care
Number analyzed (Participants) | 19 | 17
Number of infections per patient | 2 [1 to 3] | 2 [0 to 3]
Statistical Analysis 1: Comparison: Standard of Care vs NLFU and Standard of Care; Change in number of infections were not normally distributed and differences between the arms were tested using the non-parametric Mann-Whitney U test; Test type: Superiority or Other; p = 0.346, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Non-serious Adverse Events in Each Group
Description: Adverse events (AEs) were defined as any undesirable clinical occurrence in a subject whether it is thought to be related to the investigational device or not.
Time Frame: Week 5 to 13
Measure: Number; unit: Number of non-serious AEs
Arm/Group | Standard of Care | NLFU and Standard of Care
Number analyzed (Participants) | 19 | 17
Number of non-serious AEs | 70 | 59

6. Primary Outcome: Actual Change in Wound Area
Description: as for outcome 1
Time Frame: Week 5 to 13
Population: As previous
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Standard of Care | NLFU and Standard of Care
Number analyzed (Participants) | 19 | 17
cm2 | -5.3 (5.5) | -6.2 (5.5)
Statistical Analysis 1: Comparison: Standard of Care vs NLFU and Standard of Care; Test type: Superiority or Other; p = 0.618, ANCOVA; Patients' baseline (week 5) wound area was used as the covariate; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-4.7 to 2.9]

7. Secondary Outcome: Wound Recurrence Rate
Description: Patients whose wound has healed (defined as 100% epithelialisation with no scab present) before or at the end of treatment will be asked 90 days after date of healing if their wound has remained closed.
Time Frame: 90 days after time of healing
Population: Three patients healed during the study period (one NLFU+SOC patient healed after 7 weeks and one after 8 weeks of NLFU+SOC treatment, and one patient who received standard care alone healed after 4 weeks). All three of these patients remained healed 90 days after the end of their study treatment.
Measure: Number; unit: Number of wounds remained healed
Arm/Group | Standard of Care | NLFU and Standard of Care
Number analyzed (Participants) | 1 | 2
Number of wounds remained healed | 1 | 2

ADVERSE EVENTS:
Time Frame: Study period of 13 weeks
Description: Any undesirable clinical occurrence in a subject whether it is thought to be related to the NLFU or not. All subjects experiencing AEs were monitored until symptoms subside or until there is a satisfactory explanation for the changes observed. The nature of venous leg ulcers meant that AEs were common in both the SOC and NLFU groups
Arm/Group | Standard of Care | NLFU and Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 19/19 | 15/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=19) | NLFU and Standard of Care (N=17)
All adverse events (General disorders) | 19 | 15 — Any undesirable clinical occurrence in a subject whether it is thought to be related to device or not. The recording of adverse events means that specific AE terms cannot be included. See outcome relating to infection.

LIMITATIONS AND CAVEATS:
Difference in treatment frequency between the groups which could potentially bias results.

Standard deviation proved to be larger than estimated from the available literature which resulted in the study having reduced statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes